CLINICAL TRIAL: NCT01415440
Title: Examining the Effects of Stimulant Medication on Emotional Lability in Patients With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Imaging the Effects of Stimulant Medication on Emotional Lability in Patients With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Jonathan Posner, Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6235/7261R
Record Dates: First submitted 2011-07-26; First posted 2011-08-12 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Vyvanse; stimulant medication; ADD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate; Sugars

STUDY DESIGN:
Intervention Model Description: Two treatment arms plus sample of healthy controls, who were assessed at one time point
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychostimulant (Experimental): 30-70 mg capsule of Lisdexamfetamine once daily for 12 weeks
  Interventions: Drug: Lisdexamfetamine
- Placebo (Placebo Comparator): 30-70 mg capsule of placebo (sugar pill) once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine — During the first 4 weeks of treatment, the dosage of Lisdexamfetamine will be adjusted based on the patient's response to the medication. The patient will then be maintained at the lowest effective dose for the remaining 8 weeks of treatment.
  Other Names: Vyvanse
  Arms: Psychostimulant
Drug: Placebo — Placebo dosing will parallel that of Lisdexamfetamine.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The aim of this study is to examine the mechanisms by which stimulant medications reduce symptoms in patients with Attention Deficit Hyperactivity Disorder (ADHD). Using Magnetic Resonance Imaging (MRI), the investigators have found that the volumes of certain brain regions are reduced in patients with ADHD. The reduced volumes were much less pronounced if patients had been treated with stimulant medications, suggesting that stimulants may reduce the symptoms of ADHD by reversing these volume reductions. In a second and related study, the investigators found that in patients with ADHD, emotional processing was normalized when patients were taking stimulant medications. Both studies point to possible mechanisms by which stimulants are effective; however, a significant limitation of these findings is that they were derived from cross-sectional studies.

In this current study, the investigators hope to replicate these treatment effects of stimulants in a prospective, controlled manner. The investigators plan to measure ADHD symptom severity in patients before and after 12-weeks of controlled treatment with either a stimulant medication or placebo while utilizing structural and functional MRI. Combining imaging with a randomized controlled trial will allow us to better assess the effects of stimulants on brain function and structure.

DETAILED DESCRIPTION:
A cohort of 100 patients with ADHD will be recruited for a 12 week, double-blind, parallel, randomized controlled trial of Lisdexamfetamine (Vyvanse) versus placebo, with 50 patients randomized to Lisdexamfetamine and the other 50 patients to placebo. The investigators will acquire high-resolution, anatomical and functional MRI images at baseline and after 12 weeks of treatment.

In addition, 75 age- and sex-matched healthy control subjects will be imaged at baseline.

ELIGIBILITY:
Inclusion Criteria:

ADHD Participants: Meets Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD, any subtype.

Healthy Control Participants: No current DSM-IV-TR Axis I psychiatric diagnosis.

All Participants:

1. Male or female, 6 - 25 years of age, and in good physical health
2. English-speaking

Exclusion Criteria:

1. Current comorbid DSM-IV-TR Axis I psychiatric diagnosis or other symptomatic manifestations that, in the opinion of the examining physician, will contraindicate Lisdexamfetamine treatment or confound safety assessments
2. Meets DSM-IV-TR criteria for active substance abuse and/or dependence
3. Lifetime history of cocaine or stimulant abuse or dependence
4. Actively suicidal
5. Children and adolescents: Prior treatment with psychostimulants for longer than 1 month duration and/or treatment with psychostimulants within the past 4 months Adults: Treatment with psychostimulants within the past 12 months.
6. Documented allergy or intolerance to Lisdexamfetamine or other stimulant medications.
7. Taking other medications with central nervous system effects.
8. History of seizure (other than febrile seizure)
9. Diagnosis of hyperthyroidism, glaucoma, or other serious medical illness.
10. Personal or family history of medical conditions, such as cardiovascular disease, that may interfere with study participation, or for which treatment with Lisdexamfetamine may pose a risk
11. Pregnant or lactating
12. MRI contraindications such as pacemaker, braces, etc.
13. Full scale intelligence quotient (FSIQ) less than 70

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 117 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Posner, M.D, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Kessel E, Lee S, Hong S, Raffanello E, Hulvershorn LA, Margolis A, Peterson BS, Posner J. Causal effects of psychostimulants on neural connectivity: a mechanistic, randomized clinical trial. J Child Psychol Psychiatry. 2022 Nov;63(11):1381-1391. doi: 10.1111/jcpp.13585. Epub 2022 Feb 9. PMID 35141898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in 2011 and ended in 2018. Participants were primarily recruited from the community through advertisements in local newspapers and flyers posted in local establishments. Participants were also recruited from other research studies and doctor's offices.
Pre-assignment Details: 18 ADHD participants withdrew or were excluded from the study prior to randomization and thus are not included. Participants who withdrew were no longer interested in treatment or were lost to follow-up. Participants were excluded due to subthreshold ADHD symptoms, comorbid psychiatric conditions, & MRI contraindications.
Groups:
- Healthy Control: Baseline evaluation only
- ADHD - Placebo: ADHD participants randomized to receive placebo for 12 weeks of treatment
- ADHD - Vyvanse: ADHD participants randomized to receive 12 weeks of medication treatment with Vyvanse
Period: Overall Study
Arm/Group | Healthy Control | ADHD - Placebo | ADHD - Vyvanse
Started | 41 | 29 | 29
Completed | 37 | 28 | 27
Not Completed | 4 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population includes participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | ADHD - Placebo | ADHD - Vyvanse | Total
Number analyzed (Participants) | 37 | 28 | 27 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis population includes participants who completed the study.
  years | 16.54 (6.03) | 11.93 (5.72) | 12.85 (5.68) | 14.16 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 9 | 33
  Male | 22 | 19 | 18 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 21 | 6 | 9 | 36
  Race/Ethnicity: Black or African American | 6 | 11 | 4 | 21
  Race/Ethnicity: Hispanic | 7 | 7 | 10 | 24
  Race/Ethnicity: Asian or Pacific Islander | 1 | 3 | 2 | 6
  Race/Ethnicity: American Indian/Alaska Native | 0 | 0 | 0 | 0
  Race/Ethnicity: Other or Unknown | 2 | 1 | 2 | 5
Brain Structure Volume [Mean (Standard Deviation); unit: mm^3] — Population: Analysis population includes participants who completed the study.
  mm^3
    Left Hippocampal Volume | 4182.87 (418.83) | 3933.96 (433.45) | 4121.96 (392.76) | 4090.25 (424.92)
    Left Amygdala Volume | 1504.81 (217.54) | 1423.08 (199.23) | 1489.02 (235.93) | 1475.62 (218.31)
    Right Hippocampal Volume | 4288.01 (358.26) | 4011.48 (413.65) | 4185.40 (379.97) | 4174.96 (395.07)
    Right Amygdala Volume | 1695.09 (187.81) | 1577.34 (204.15) | 1665.87 (234.17) | 1651.16 (210.79)

OUTCOME MEASURES:

1. Primary Outcome: Brain Structure Volume
Description: Brain structure volume measured in mm^3
Time Frame: 12 weeks
Population: ADHD participants who completed 12 weeks of treatment.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | ADHD - Placebo | ADHD - Vyvanse
Number analyzed (Participants) | 27 | 28
mm^3
  Left Hippocampal Volume | 3909.85 (535.35) | 4069.72 (426.46)
  Left Amygdala Volume | 1431.31 (245.40) | 1485.05 (235.17)
  Right Hippocampal Volume | 4048.10 (454.37) | 4206.41 (413.38)
  Right Amygdala Volume | 1573.57 (240.03) | 1641.88 (207.45)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, an average of 12 weeks.
Description: Adverse events were routinely collected from ADHD participants receiving treatment using the Pittsburgh Side Effects Rating Scale. A physician met with participants in person approximately once per week during treatment. The physician was also available by phone between visits.
Arm/Group | Healthy Control | ADHD - Placebo | ADHD - Vyvanse
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/41 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT01415440/Prot_SAP_000.pdf